CLINICAL TRIAL: NCT02913287
Title: A Randomised, Double-blind, Placebo-controlled Study of the Cognitive-Enhancing Potential of Seaweed-Derived Mineral-Rich Nutraceuticals (a Combination of Aquamin F and Aquamin MG)
Brief Title: Seaweed-Derived Mineral-Rich Nutraceuticals in Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YN001
Record Dates: First submitted 2016-09-19; First posted 2016-09-23 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Cognition
MeSH Terms: interventions — Aquamin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Other: Maltodextrin Placebo
- Aquamin/Aquamin MG (Experimental): Aquamin/Aquamin MG mix
  Interventions: Dietary Supplement: Aquamin/Aquamin MG

INTERVENTIONS:
Dietary Supplement: Aquamin/Aquamin MG — Marine-based nutraceutical
  Arms: Aquamin/Aquamin MG
Other: Maltodextrin Placebo — Maltodextrin Placebo
  Arms: Placebo

SUMMARY:
The aim of the overall project is to investigate the potential of a combination of commercially available nutraceuticals produced by Marigot Ltd (natural seawater derived mineral-rich AquaminMG and seaweed-derived mineral-rich food supplement AquaminTM (FDA GRAS 000028) isolated from Lithothamnion species), as safe and effective supplements to promote cognition in the aged brain.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrolment into the study, subjects must;

1. Be able to give written informed consent.
2. Be between 65 and 85 years of age (elderly cohort).
3. If female, must be non-pregnant.
4. Be in generally good health as determined by the investigator.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the below criteria;

1. Are less than 65 and greater than 85 years of age (elderly cohort).
2. Are pregnant females.
3. Are currently taking calcium/magnesium supplements, or have taken them in the past 14 days.
4. Have a significant acute or chronic co-existing illness (cardiovascular, gastrointestinal, endocrinological, immunological, metabolic or any condition which contraindicates, in the investigators judgement, entry to the study).
5. Have a score of <22 in the Montreal Cognitive Assessment (MoCA) (elderly cohort) and have no subjective memory impairment.
6. Have a history of renal failure or renal disease, or eGFR creatinine levels below 30ml/min.
7. Have diagnosis of significant low or high calcium or magnesium levels.
8. Have a condition or are taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; to include misoprostrol, polystyrene sulfonate, Riociguat and vitamin/mineral supplements, probiotics or herbal remedies.
9. Are individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
10. Are receiving treatment involving experimental drugs.
11. Have been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.
12. Have a malignant disease or any concomitant end-stage organ disease.
13. Have a psychiatric illness which contraindicates entry to the study.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Cognition as measured using CANTAB tests | On study completion, after each individual completes 12 weeks of supplement

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Nolan, Principal Investigator — University College Cork
Locations (1):
- University College Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided